CLINICAL TRIAL: NCT04709536
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study Evaluating the Efficacy and Safety of IBI306 in Patients With Hypercholesterolemia in China (CREDIT-4)
Brief Title: A Study of IBI306 in Participants With Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBI306B201
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI306 (Experimental): IBI306 administered subcutaneously (SC)
  Interventions: Drug: IBI306
- Placebo (Placebo Comparator): administered subcutaneously (SC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IBI306 — Recombinant humanized Anti- PCSK9 monoclonal antibody, administered SC from BL to week 24
  Arms: IBI306
Drug: Placebo — Recombinant humanized Anti- PCSK9 monoclonal antibody, administered SC from BL to week 24
  Arms: Placebo

SUMMARY:
This study is designed for multi-center, double-blind, randomized, placebo-controlled phase III trial to evaluate the safety and tolerability of subcutaneous injection of IBI306 in hypercholesterolemia patients.

ELIGIBILITY:
Inclusion criteria

1. Males and females ≥ 18 to ≤ 75 years of age
2. Diagnosis of hypercholesterolemia
3. LDL cholesterol ≥ 70 mg/dl (1.8mmol/L)
4. Very high or high cardiovascular risk
5. TG≤500 mg/dL(5.64 mmol/L)

Exclusion criteria

1. Uncontrolled hypertension
2. Uncontrolled hyperthyroidism or hypothyroidism
3. Severe renal dysfunction
4. Known sensitivity to any of the products to be administered during dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
1. Mean percent change from baseline in low-density lipoprotein cholesterol (LDL-C) at weeks 12 | Baseline to week12

SECONDARY OUTCOMES:
The percent of subjects with LDL-C reduction no less than 50% from baseline | Baseline to week24
The percent of subjects with LDL-C<70mg/dL(1.8 mmol/L) | Baseline to week24
The percent change in Lp(a),ApoB, non-HDL-c, ApoB/ApoA1 from baseline | Baseline to week24

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

REFERENCES:
- [Derived] Qi L, Liu D, Qu Y, Chen B, Meng H, Zhu L, Li L, Wang S, Liu C, Zheng G, Lian Q, Yin G, Lv L, Lu D, Chen X, Xue F, An P, Li H, Deng H, Li L, Qian L, Huo Y. Tafolecimab in Chinese Patients With Hypercholesterolemia (CREDIT-4): A Randomized, Double-Blind, Placebo-Controlled Phase 3 Trial. JACC Asia. 2023 Jul 11;3(4):636-645. doi: 10.1016/j.jacasi.2023.04.011. eCollection 2023 Aug. PMID 37614541